CLINICAL TRIAL: NCT03542435
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of SXC 2023 When Administered Orally to Healthy Adult Subjects
Brief Title: Randomized, Double-Blind, Placebo-Controlled, MAD Study to Assess the Safety, Tolerability, and Pharmacokinetics of SXC 2023
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Promentis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-104
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SXC-2023 (Experimental): Dose Escalation
  Interventions: Drug: SXC-2023
- Placebo (Placebo Comparator): Dose Escalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SXC-2023 — Oral capsule
  Arms: SXC-2023
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple ascending dose study conducted at one study center in the United States. Safety and tolerability will be assessed throughout the study and serial blood samples and urine samples will be collected for the safety and pharmacokinetic assessment of SXC-2023.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female, 18 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose and throughout the study.
3. BMI ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant screening results.
5. For a female of childbearing potential: either be sexually inactive (abstinent as a life style) for 28 days prior to the first dosing and throughout the study or be using acceptable birth control methods:
6. Female of non childbearing potential: must have undergone sterilization procedures, at least 6 months prior to the first dose
7. Non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug/placebo.
8. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated
2. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
3. History or presence of alcoholism or drug abuse within the past 2 years
4. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
5. Females with a positive pregnancy test or is lactating.
6. Positive urine cotinine at screening.
7. Positive urine drug or alcohol results at screening
8. Any significant finding on the Columbia Suicidal Severity Rating Scale (C-SSRS)
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
10. Unable to refrain from or anticipates the use of any drug (e.g. prescription, recreational, etc.)
11. Donation of blood or significant blood loss within 56 days prior to the first dose.
12. Plasma donation within 7 days prior to the first dose.
13. Participation in another clinical study within 30 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | 18 days
  Treatment related adverse events as a measure of safety and tolerability of SXC-2023 following multiple ascending doses

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: Cmax | Up to 96 hr post dose
  Peak plasma concentration
Pharmacokinetic Assessments: Tmax | Up to 96 hr post dose
  Time to peak plasma concentration
Pharmacokinetic Assessments: AUC | Up to 96 hr post dose
  Area under the plasma concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Cotter, Study Director — Promentis Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No